CLINICAL TRIAL: NCT00331708
Title: An Open-label in Vivo Drug Study to Evaluate Artesunate Plus Sulfadoxine-pyrimethamine (ASSP) Pharmacokinetics, Therapeutic Efficacy, Gametocyte Carriage and Birth Outcomes in Pregnant Women With Uncomplicated Falciparum Malaria
Brief Title: Artesunate Plus Sulfadoxine-pyrimethamine Pharmacokinetics, Efficacy, Gametocytes Carriage and Birth Outcomes in Pregnant Women With Malaria
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of suitable participants
Sponsor: Professor Karen I Barnes (Other)
Collaborators: Global Fund (Other); Medical Research Council, South Africa (Other)
Responsible Party: Sponsor-Investigator, Professor Karen I Barnes, Professor, Clinical Pharmacology, University of Cape Town
Organization: University of Cape Town (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEACAT2.1
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Malaria
Keywords: Malaria; Efficacy; Pharmacokinetic; Gametocyte; Molecular markers; Sulfadoxine-pyrimethamine; Artesunate; Artemisinin
MeSH Terms: conditions — Malaria | interventions — Artesunate; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Artesunate plus sulphadoxine-pyrimethamine (Experimental)
  Interventions: Drug: Artesunate plus sulfadoxine-pyrimethamine

INTERVENTIONS:
Drug: Artesunate plus sulfadoxine-pyrimethamine

SUMMARY:
The main purpose of this study is to compare the drug levels of artesunate and sulfadoxine-pyrimethamine found in pregnant women with malaria to those drug levels found in non-pregnant women from other studies. In addition the efficacy and safety of the study drugs will be determined for pregnant women and their babies.

DETAILED DESCRIPTION:
The resistance of Plasmodium falciparum to anti-malarial drugs is a serious impediment to the control of malaria, and this poses a particular problem for the treatment of pregnant women, a group especially vulnerable to malaria; pregnancy increases the risk of disease progression and complications with up to a 10-fold increase in the malaria case fatality rate in areas of low transmission. As falciparum parasites can sequester in the placenta, pregnant women have been shown to develop recrudescence up to 85 days after quinine treatment, and are at increased risk of gametocyte carriage. Artemisinin-based combination therapies have been shown to improve cure rates and to delay antimalarial resistance. In humans the efficacy and safety of artesunate in the treatment of malaria in pregnancy has been studied in over 1000 women in which no evidence of foetal harm was demonstrated. Quinine is the only alternative currently available in Mozambique for treating malaria in pregnancy however there is relatively little data available on its efficacy or safety. There is no published information on the pharmacokinetics of SP in pregnancy, however data show a marked reduction in bioavailability of artesunate and its active metabolite, dihydroartemisinin. Thus, we cannot be confident that the standard dosage regimens of SP and of artesunate are optimal for the treatment of acute uncomplicated malaria in pregnancy or whether altered pharmacokinetics is contributing to the SP-treatment failures observed in pregnancy. This study creates the opportunity to study whether the pharmacokinetic properties of SP and artesunate are altered by physiological changes that occur during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female, older than 18 years, > 35kg.
* Gestational age > 16 weeks (fundal height > 16cm) and below 36 weeks gestation.
* Diagnoses of uncomplicated acute P. falciparum malaria parasitaemia of up to 250 000 asexual parasites/ul blood with axillary temperature of greater than or equal to 37.5°C or history of fever (defined as fever within the previous 24 hours).
* Documented written informed consent.
* Lives close enough to the study site for reliable follow up and is willing to attend ANC and follow-up visits regularly.
* Is willing to stop taking folate for 7 days if applicable.

Exclusion Criteria:

* Has received anti-malarial treatment in the past 7 days.
* Severely ill (based on WHO Criteria for severe malaria ) or if patient is considered, in the opinion of the investigator or designee, to have moderately severe malaria (e.g. prostrate, repeated vomiting, dehydrated) or other danger signs (Appendix 2).
* Known hepatic or renal impairment
* Has received chloramphenicol or tetracyclines (including doxycycline) in the past 7 days or is likely to require these during the study period.
* History of G6PD deficiency.
* Has a history of allergy to any of the study drugs (including other sulphonamides e.g. cotrimoxazole, or other artemisinin derivatives e.g. co-artemether).
* Serious underlying disease that in the opinion of the clinic team and/or Principal Investigator would make the patient unsuitable for the study in terms of their safety or study analysis.
* Imminent delivery expected.
* Prior inclusion in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters by measurement of whole blood levels of sulfadoxine and pyrimethamine and plasma levels of artesunate and its active metabolite dihydroartemisinin to determine Cmax, Tmax, AUC, half life, volume of distribution and clearance
Correlation of treatment outcome with pharmacokinetic parameters and pregnancy status.

SECONDARY OUTCOMES:
Association of gametocyte carriage with pregnancy status
Correlation of frequency of DHFR mutations at codons 108, 51, 59 (164) and DHPS mutations at codons 436, 437, 540 and 581 in maternal and placental samples with treatment outcome
Birth outcomes in terms of congenital abnormalities, spontaneous abortions, still births and neonatal deaths, gestational age and birth weight, placental weight, newborn head circumference
Risk of harm by describing adverse events and their causality assessments, neurodevelopmental assessment of infants and changes in full blood count (or haemoglobin), glucose, bilirubin, creatinine, urea and ALT
Capacity building by describing the training and development of study teams and their subsequent skills attained.

CONTACTS AND LOCATIONS:
Overall Officials: Karen I Barnes, MBChB, Principal Investigator — University of Cape Town
Locations (1):
- Ndlavela Health Centre, Ndlavela, Maputo, Mozambique